CLINICAL TRIAL: NCT04651517
Title: Pilot Study of the XACT Robotics ACE System for Image Guided Percutaneous Procedures in the Lung
Brief Title: Pilot Study of the ACE System in Lung Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xact Robotics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLIN-LUNG-01-2020
Record Dates: First submitted 2020-11-17; First posted 2020-12-03 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Intervention Model Description: Subjects 18 years of age or older who are undergoing CT guided, minimally invasive percutaneous procedures of the lung.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Study arm (Experimental): Subjects undergoing procedures with the XACT ACE Robotic system.
  Interventions: Device: XACT ACE Robotics study arm

INTERVENTIONS:
Device: XACT ACE Robotics study arm — Subjects will undergo lung procedures with the physician utilizing the XACT ACE Robotic System.

SUMMARY:
To evaluate the XACT ACE Robotic System in lung procedures.

DETAILED DESCRIPTION:
The XACT ACE Robotic System is a user-controlled positioning system intended to assist in the planning and advancement of an instrument during Computed Tomography (CT) guided percutaneous lung procedures. The system is used for trajectory planning and is intended to assist the physician in the positioning of an instrument, such as a needle, where CT imaging is used for target trajectory planning and intraoperative tracking. This study will evaluate safety and accuracy of the XACT ACE Robotic System in subjects undergoing CT guided, minimally invasive percutaneous procedures of the lung in the interventional radiology suite.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age
2. Subjects undergoing CT-guided, minimally invasive percutaneous lung procedures in the interventional radiology suite, e.g., core biopsy, fine needle aspiration (FNA), tumor ablation, etc.
3. Following planning and registration CT scans, subject is found eligible to undergo CT-guided, minimally invasive percutaneous procedure
4. Subject is willing to sign informed consent
5. Subject is capable of adhering to study procedures

Exclusion Criteria:

1. Subjects in whom the target is within 1 cm of a major blood vessel, major nerve or heart
2. Subject with significant coagulopathy
3. Subject with preexisting or unstable medical condition(s), which in the opinion of the investigator, might interfere with the conduct of the study
4. Subjects who are pregnant or nursing
5. Following planning and registration CT scans, required clinical trajectory to target is beyond system workspace limits (e.g., entry angle is too sharp)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 30 days
  Incidence, severity, and frequency of adverse events and device-related adverse events

SECONDARY OUTCOMES:
Secondary Performance Evaluation - Clinical Accuracy | 1 hour
  Percent of procedures in which the needle reached the pre-defined target based on the physician's determination and CT imaging confirmation (clinical accuracy)
Secondary Performance Evaluation - System Accuracy | 1 hour
  The measured distance from the tip of the needle/tool to the target location at the end of the needle/tip insertion.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Flacke, MD, Principal Investigator — Lahey Hospital & Medical Center
Locations (1):
- Lahey Hospital and Medical Center, Burlington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No